CLINICAL TRIAL: NCT03093610
Title: Evaluation of Fluid Output Threshold for Safe Chest Tube Removal - A Potential Way to Decrease Length of Stay in Hospital and to Improve Postoperative Care After Lung Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14032017
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pleural Effusion Recurrence; Pulmonary Resection; Chest Tube Management

STUDY DESIGN:
Intervention Model Description: Group 1: Removal of the chest tube after air leakage has ceased and fluid Drainage is < 200ml/24h Group 2: Removal of the chest tube after air leakage has ceased and fluid Drainage is < 5ml/kg/24h
Who Masked: Care Provider
Masking Description: The operating surgeon does not know to which group the Patient will be attributed to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional (Active Comparator): The chest tube in the traditional Group will be managed according to the current Guidelines of the investigators' department.
  Interventions: Procedure: Traditional
- Test group (Active Comparator): The chest tube in the "Test Group" will constitute the experimental Group. The chest tube will be removed when the fluid production over 24h has reached a weight related threshold.
  Interventions: Procedure: Test

INTERVENTIONS:
Procedure: Traditional — Removal of the chest tube after air leakage has ceased and fluid drainage is 200ml/24h or less.
  Arms: Traditional
Procedure: Test — Removal of the chest tube after air leakage has ceased and fluid drainage is 5ml/kg/24h or less.
  Arms: Test group

SUMMARY:
Previous studies have shown that the removal of the chest tube after lung surgery significantly improves pain symptoms and lung function. The criteria for chest tube removal still remain vague in modern thoracic surgery and rely on personal experience instead of evidence-based criteria. Every hospital has its own traditional standard fluid threshold and believes in that without adapting and comparing it not even after introduction of newer and more minimal-invasive operation technique. According to literature the traditional fluid threshold is varying from 100 to 500 or even more millilitre in 24 hours. Since pleural fluid resorption is proportional to body weight the investigators believe that a body weight related approach of chest tube management would improve safety and would allow an earlier chest tube removal without a higher rate of complication. In this way the investigators believe in improving pain management and in achieving earlier discharge of the patient.

ELIGIBILITY:
Inclusion criteria:

* Lobectomy/ Bilobectomy
* Segmentectomy
* Signed consent
* Age of majority

Exclusion criteria:

* Pneumonectomy
* Atypical resections
* Empyema
* Pleural effusion (not related to surgery)
* Pleurodesis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Number of recurrent pleural effusions after chest tube removal | up to 6 weeks postoperative
  Evaluation of recurrent pleural effusion after chest tube removal
Pain scores (VAS-Score) | postoperative Period until 3 hours after Chest tube removal
  Evaluation of Pain Scores after Chest tube removal
Time Point of chest tube removal | Postoperative, expected to be up to 1 week after surgery
  postoperative day of chest tube removal

SECONDARY OUTCOMES:
Patient discharge | At time of discharge, on average 4-7 days
  Time Point of Patient discharge

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dorn, Study Director — Chief, Department of General Thoracic Surgery, Bern University Hospital
Locations (1):
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared, All participant Data will be encrypted

REFERENCES:
- [Background] Bjerregaard LS, Jensen K, Petersen RH, Hansen HJ. Early chest tube removal after video-assisted thoracic surgery lobectomy with serous fluid production up to 500 ml/day. Eur J Cardiothorac Surg. 2014 Feb;45(2):241-6. doi: 10.1093/ejcts/ezt376. Epub 2013 Jul 19. PMID 23872457
- [Background] Xie HY, Xu K, Tang JX, Bian W, Ma HT, Zhao J, Ni B. A prospective randomized, controlled trial deems a drainage of 300 ml/day safe before removal of the last chest drain after video-assisted thoracoscopic surgery lobectomy. Interact Cardiovasc Thorac Surg. 2015 Aug;21(2):200-5. doi: 10.1093/icvts/ivv115. Epub 2015 May 15. PMID 25979532
- [Background] Zhang Y, Li H, Hu B, Li T, Miao JB, You B, Fu YL, Zhang WQ. A prospective randomized single-blind control study of volume threshold for chest tube removal following lobectomy. World J Surg. 2014 Jan;38(1):60-7. doi: 10.1007/s00268-013-2271-7. PMID 24158313
- [Background] Cerfolio RJ, Bryant AS. Results of a prospective algorithm to remove chest tubes after pulmonary resection with high output. J Thorac Cardiovasc Surg. 2008 Feb;135(2):269-73. doi: 10.1016/j.jtcvs.2007.08.066. PMID 18242249
- [Background] Younes RN, Gross JL, Aguiar S, Haddad FJ, Deheinzelin D. When to remove a chest tube? A randomized study with subsequent prospective consecutive validation. J Am Coll Surg. 2002 Nov;195(5):658-62. doi: 10.1016/s1072-7515(02)01332-7. PMID 12437253
- [Background] Irshad K, Feldman LS, Chu VF, Dorval JF, Baslaim G, Morin JE. Causes of increased length of hospitalization on a general thoracic surgery service: a prospective observational study. Can J Surg. 2002 Aug;45(4):264-8. PMID 12174980
- [Background] Refai M, Brunelli A, Salati M, Xiume F, Pompili C, Sabbatini A. The impact of chest tube removal on pain and pulmonary function after pulmonary resection. Eur J Cardiothorac Surg. 2012 Apr;41(4):820-2; discussion 823. doi: 10.1093/ejcts/ezr126. Epub 2011 Dec 21. PMID 22219425
- [Background] Mueller XM, Tinguely F, Tevaearai HT, Ravussin P, Stumpe F, von Segesser LK. Impact of duration of chest tube drainage on pain after cardiac surgery. Eur J Cardiothorac Surg. 2000 Nov;18(5):570-4. doi: 10.1016/s1010-7940(00)00515-7. PMID 11053819
- [Background] STEWART PB. The rate of formation and lymphatic removal of fluid in pleural effusions. J Clin Invest. 1963 Feb;42(2):258-62. doi: 10.1172/JCI104712. No abstract available. PMID 13984113